CLINICAL TRIAL: NCT00401609
Title: Evaluation of Activity and Toxicity of Polychemotherapy With 2-drug Combinations Containing Gemcitabine as First Line Treatment of Elderly Patients With Small Cell Lung Cancer
Brief Title: G-Step: Gemcitabine Based Small-cell Lung Cancer Treatment in Elderly Patients
Acronym: G-Step
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Francesco Perrone, NCI Naples
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G-Step
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Small Cell Lung Cancer
Keywords: elderly
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Gemcitabine; Vinorelbine; Cisplatin; Etoposide; Carboplatin

INTERVENTIONS:
Drug: gemcitabine
Drug: vinorelbine
Drug: cisplatin
Drug: etoposide
Drug: carboplatin

SUMMARY:
The purpose of this study is to describe the activity and toxicity of gemcitabine combined with four different drugs (carboplatin or cisplatin or etoposide or vinorelbine) as first line treatment of elderly patients with extensive small cell lung cancer.

DETAILED DESCRIPTION:
Four treatment arms are planned.

* GEMVIN: gemcitabine 1000 mg/m2 and vinorelbine 25 mg/m2 on days 1 & 8, every 21 days
* GEMCAR: gemcitabine 1000 on days 1 & 8 and carboplatin AUC 3.5 or 4 or 4.5 on day 1, every 21 days
* GEMCIS: gemcitabine 1000 mg/m2 on days 1 & 8 and cisplatin 50 or 60 or 70 mg/m2 on day 1, every 21 days
* GEMETO: gemcitabine 1000 mg/m2 on days 1 & 8 and etoposide 60 or 70 or 80 mg/m2 on days 1,2,3 every 21 days

For the study of the GEMVIN combination a two-stage minimax flexible design will be applied. For the remaining 3 combinations (GEMCAR, GEMCIS, GEMETO) a phase 1/2 design aimed at looking for optimal dose within a Bayesian framework will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of SCLC
* Extensive disease
* Measurable disease
* Performance Status (ECOG) < o = 2
* Age > o = 70 years.
* Written informed consent.

Exclusion Criteria:

* Previous chemotherapy.
* Previous or concomitant malignancies (with the exception of adequately treated non melanomatous skin cancer or carcinoma in situ of the cervix)
* •Neutrophils<2.000/mm3;platelets<100.000/mm3; hemoglobin < 10 g/dl
* Creatinine > 1.5 time the upper limit
* AST, ALT > 2.5 times and/or bilirubin > 1.5 time the upper limit of normal if liver metastases are absent or AST, ALT ³5 times and bilirubin > 3 times the upper limit of normal if liver metastases are present
* Symptomatic brain metastases

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 85
Dates: Start 2000-11; Primary Completion 2007-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
to evaluate activity and toxicity of GEMVIN combination
to identify optimal dose of GEMETO, GEMCAR, and GEMCIS combinations
to evaluate activity and toxicity of GEMETO, GEMCAR, and GEMCIS combinations

SECONDARY OUTCOMES:
treatment impact on patient quality of life
prognostic value of ADL and IADL multidimensional geriatric evaluation scales
clinical variables predictive of response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Gridelli, M.D., Principal Investigator — San Giuseppe Moscati Hospital, Avellino, Italy; Francesco Perrone, M.D., Ph.D., Principal Investigator — National Cancer Institute Naples, Italy
Locations (21):
- Italy (21):
  - Azienda Ospedaliera S. Giuseppe Moscati, U.O. di Oncologia Medica, Monteforte Irpino, AV
  - IRCCS Oncologico Bari, Oncologia Medica, Bari, BA
  - Ospedale A. Cardarelli, Campobasso, CB
  - Ospedale Mariano Santo, U.O. di Oncologia Medica, Cosenza, CS
  - Ospedale Umberto di Frosinone, Frosinone, FR
  - Umberto I SS. Trinita' Ospedale, Frosinone, FR
  - Ospedale San Martino, Genova, GE
  - Ospedale Serbelloni, Gorgonzola, MI
  - Policlinico Universitario P. Giaccone, Palermo, PA
  - Ospedale La ferla, Palermo, PA
  - Policlinico Giaccone, Palermo, PA
  - Istituto Oncologico Veneto, Padua, PD
  - Istituto Regina Elena, Divisione di Oncologia Medica, Roma, Roma
  - Ospedale S. Giovanni Calibita Fatebenefratelli, Roma, Roma
  - Ospedale Civile, Polla, SA
  - Divisione di Oncologia Medica, U.S.L.L. 13, Noale, VE
  - Ospedale L. Sacco, Milan
  - Istituto Nazionale dei Tumori , Divisione di Oncologia Medica B, Napoli
  - Ospedale Monaldi, Napoli
  - Azienda Sanitaria Locale 2, Pozzuoli
  - Ospedale San Camillo - Forlanini, Rome

REFERENCES:
- [Result] Gridelli C, Gallo C, Morabito A, Iaffaioli RV, Favaretto A, Isa L, Barbera S, Gamucci T, Ceribelli A, Filipazzi V, Maione P, Rossi A, Barletta E, Signoriello S, De Maio E, Piccirillo MC, Di Maio M, Rocco G, Vecchione A, Perrone F; G-STEP Investigators. Phase I-II trial of gemcitabine-based first-line chemotherapies for small cell lung cancer in elderly patients with performance status 0-2: the G-STEP trial. J Thorac Oncol. 2012 Jan;7(1):233-42. doi: 10.1097/JTO.0b013e318233d6c2. PMID 22031232